CLINICAL TRIAL: NCT01606072
Title: Perioperative Administration of Desmopressin to Subjects With Breast Cancer: A Phase IIa, Dose-Escalation Study
Brief Title: Perioperative Use of Desmopressin (DDAVP) in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DDAVP
Record Dates: First submitted 2012-05-11; First posted 2012-05-25 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer
Keywords: DDAVP
MeSH Terms: conditions — Breast Neoplasms | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Desmopressin (Experimental)
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — 20 patients in 5 groups 4 each, advancing progressively to each dose level.

SUMMARY:
The propose for this study is to evaluate the safety and tolerability of desmopressin when administered perioperatively to patients with breast cancer undergoing surgery as first treatment, and select the optimum dose for the clinical development of the product.

DETAILED DESCRIPTION:
Breast cancer is one of the most commonly diagnosed malignancies among women, and its mortality is related to the capacity of tumor cells to invade and produce metastases. It is postulated that tumor manipulation during surgery results in the release of tumor cells into circulation or the lymphatic system, and that these released cells survive due to aggregation among them or with platelets through the formation of a fibrin layer on the embolus. Tumor cells surviving transportation through circulation will join blood vessels and invade vascular walls, forming metastases. The interruption of this process might reduce survival of tumor cells and thus the formation of metastases from breast cancer cells in the lungs or other tissues.

ELIGIBILITY:
Inclusion Criteria:

* a. Female subjects from 21 to 60 years of age, who have voluntarily signed the informed consent form.

  b. Histological/cytological diagnosis of breast carcinoma obtained at least 21 days before inclusion into the study.

  c. Candidate for radical mastectomy and requiring resection of axillary lymph nodes or sentinel node.

  d. In case of women of childbearing potential, an adequate birth control method (intrauterine device, barrier methods, or tubal ligation) should be used throughout the study. Post-menopausal women should have menopause confirmed by biochemical parameters.

  e. Adequate organic function, defined by the following parameters:
  * Electrocardiogram (ECG) with no significant anomalies, performed within 14 days prior to surgery.
  * The following laboratory results, obtained 7 days before surgery:
  * Hemoglobin ≥ 11 g/dL
  * Total white blood cell count ≥ 4,000/mm3
  * Total neutrophil count 1,500/mm3
  * Platelet count within normal limits
  * Total bilirubin ≤1.5 x UNL or 2.5 x UNL in case of hepatic metastasis
  * Transaminases ALT/GPT and AST/GOT ≤ 1.5 x UNL
  * Creatinine clearance >50 mg/dL
  * CT scan with oral and endovenous contrast* of chest, pelvis, and abdomen, and bone scan, conducted within 28 days prior to surgery. Images taken not longer than 90 days before surgery are also acceptable.

    * In case contrast is contraindicated, CT with no contrast or MRI will be performed.

      f. Subject with performance status (ECOG) = 0.

Exclusion Criteria:

* a. Synchronic bilateral breast cancer. b. Symptoms of metastasis or evidence of metastasis from images: chest spiral CT scan, abdomen/pelvis spiral CT scan, brain spiral CT/MRI (in case of brain metastasis signs), and bone scan.

  c. The patient is pregnant or breastfeeding. d. The patient is presently using hormonal contraceptives or under hormonal treatment. She would be eligible if oral contraceptives were discontinued or if the hormonal treatment finished 30 days before surgery and the patient agreed to use another contraceptive method.

  e. Patients with a history or presence of congestive heart failure, blood hypertension, angina pectoris or heart arrhythmia, thromboembolic disease, diabetes type I or II, or any underlying coronaropathy detected in pre-surgical evaluations.

  f. Mentally-impaired patients. g. Patients with known hypersensitivity to DDAVP or vasopressin, o with severe von Willebrand's disease (VWD), defined by a VWF activity <10%IU/dL, or type 2B VWD, defined by an increased ristocetin-induced platelet aggregation (RIPA) at low concentrations of ristocetin or with hemophilia.

  h. Patients with a history of seizures. i. Patients with renal impairment (creatinine clearance < 50 mL/min calculated by the Cockcroft-Gault formula), hyponatremia or with a history of hyponatremia.

  j. Patients with syndrome of inadequate secretion of antidiuretic hormone. k. Patients with positive serology for the hepatitis B or C virus and/or HIV. l. Patients with known hepatic disease (diagnosed cirrhosis, hepatic enzymes (GOT/GPT) > 1.5 x UNL, Total bilirubin > 1.5 x UNL).

  m. Patients with active infections. n. Patients with other malignant diseases, with the exception of, non-melanoma skin cancer, or cervix cancer in situ, or any other tumor that has received adequate treatment and shows a disease-free time ≥ 5 years.

  o. Patients participating in another clinical study or cases in which less than 4 weeks have elapsed since participation in another clinical study.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Selection of the higher safe dose level for ensuing clinical trials | Up to 2 years
  One of the three dose levels assessed in this study will be selected for further clinical testing in adults: 0,50 mg, 1,0 mg, 1,25 mg, 1,5 mg or 2,0 mg.

SECONDARY OUTCOMES:
Evidence of V2 Receptor Expression | Baseline
Evidence of CTC (CIRCULATING TUMOR CELLS) | Baseline
Evidence of Von Willebrand factor antigen (VWF:Ag) | Baseline
Evidence of CTC (circulating tumor cells) | 30 minutes pre surgery and 24 hours post the surgery
Evidence of CTC (circulating tumor cells) | 2 Weeks
Evidence of CTC (circulating tumor cells) | 1 Month
Evidence of CTC (circulating tumor cells) | 3 Months
Evidence of CTC (circulating tumor cells) | 6 Months
Evidence of CTC (circulating tumor cells) | 12 Months
Evidence of Von Willebrand factor antigen (VWF:Ag) | 120 minutes post the surgery
Evidence of VWF activity (ristocetin cofactor, VWF:RCo) | baseline
Evidence of VWF activity (ristocetin cofactor, VWF:RCo) | 120 minutes post the surgery
Evidence of FVIII coagulant activity (FVIII:C) | baseline
Evidence of FVIII coagulant activity (FVIII:C) | 120 minutes post the surgery
Evidence of euglobulin lysis time | baseline
Evidence of euglobulin lysis time | 120 minutes post the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dra. Ruth Weinberg, Principal Investigator — Hospital Interzonal General De Agudos Eva Peron
Locations (1):
- Hospital Interzonal General De Agudos EvaPeron, Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Result] Weinberg RS, Grecco MO, Ferro GS, Seigelshifer DJ, Perroni NV, Terrier FJ, Sanchez-Luceros A, Maronna E, Sanchez-Marull R, Frahm I, Guthmann MD, Di Leo D, Spitzer E, Ciccia GN, Garona J, Pifano M, Torbidoni AV, Gomez DE, Ripoll GV, Gomez RE, Demarco IA, Alonso DF. A phase II dose-escalation trial of perioperative desmopressin (1-desamino-8-d-arginine vasopressin) in breast cancer patients. Springerplus. 2015 Aug 19;4:428. doi: 10.1186/s40064-015-1217-y. eCollection 2015. PMID 26306290